CLINICAL TRIAL: NCT05459727
Title: Effects of Non-surgical Periodontal Therapy on Cardiovascular Risk in People at Risk of Cardiovascular Disease
Brief Title: Effects of Non-surgical Periodontal Therapy on Cardiovascular Risk
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Nanfang Hospital, Southern Medical University (Other)
Collaborators: Southern Medical University, China (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: NFEC-2022-243
Record Dates: First submitted 2022-07-05; First posted 2022-07-15 (Actual); Last update posted 2022-07-15 (Actual); Status verified 2022-05

CONDITIONS: Cardiovascular Diseases; Periodontitis
Keywords: Periodontitis; Non-surgical Periodontal Therapy; Cardiovascular risk
MeSH Terms: conditions — Cardiovascular Diseases; Periodontitis

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Masking Description: Due to the characteristics of the intervention in this trial, it would be impossible to blind the enrolled participants. However, the investigators and outcomes assessors will be blinded. Allocation to arms will be concealed in an envelope and revealed to the stomatologist and patient before delivering the first treatment. Other investigators like outcomes assessors and staff involved in the data collection and analyses will be masked.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention arm (Experimental): 1. Basic oral hygiene instructions.
  2. Full-mouth subgingival scaling and root planing under local anesthesia.
  3. Additional full-mouth subgingival scaling and root planing under local anesthesia every 3 months during the follow-up period if necessary.
  Interventions: Procedure: Non-surgical periodontal therapy
- Control arm (Placebo Comparator): 1. Basic oral hygiene instructions.
  2. Full-mouth supragingival ultrasonic scaling.
  Interventions: Procedure: Control periodontal treatment

INTERVENTIONS:
Procedure: Non-surgical periodontal therapy — Non-surgical periodontal therapy includes basic oral hygiene instructions and full-mouth subgingival scaling and root planing under local anesthesia.
  Arms: Intervention arm
Procedure: Control periodontal treatment — Control periodontal treatment includes basic oral hygiene instructions and full-mouth supragingival ultrasonic scaling.
  Arms: Control arm

SUMMARY:
This study is to evaluate whether non-surgical periodontal therapy can help to control the cardiovascular risk among patients with moderate/severe periodontitis and at risk of cardiovascular disease.

DETAILED DESCRIPTION:
Previous studies showed that the treatment of periodontitis can partially improve the control of risk factors of cardiovascular disease (e.g. blood pressure, interleukin 6), whereas the evidence is still limited. Moreover, there is currently no study reporting the impact of periodontal treatment on the overall risk of cardiovascular disease. The prevalence of periodontitis in China was 62.4%. In clinical practice, a large number of patients with moderate/severe periodontitis and at risk of cardiovascular disease seek medical advice. However, the existing guidelines lack relevant recommendations. Therefore, this study intends to evaluate whether non-surgical periodontal therapy can help to control cardiovascular risk.

376 patients with moderate/severe periodontitis and at risk of cardiovascular disease will be randomized. Those randomized to the intervention arm will receive non-surgical periodontal therapy which includes full-mouth subgingival scaling and root planing. Those randomized to the control arm will receive supragingival ultrasonic scaling. All patients were given instructions on basic oral hygiene.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years;
* At risk of cardiovascular disease (defined as "Framingham Score" predicted 10-year risk of cardiovascular disease ≥ 20%);
* Moderate//severe periodontitis;

Exclusion Criteria:

* Cardiovascular diseases at baseline (coronary heart disease, stroke and peripheral artery disease);
* Received periodontal treatment within the past 6 months;
* Pregnant or lactating females;
* Non residents of Guangzhou and its surrounding cities or expected to leave Guangzhou or its surrounding cities within 1 year;
* Malignant tumors or other end-stage diseases with life expectancy less than 1 year;
* End-stage renal disease;
* Patients with high bleeding risk, high blood pressures or other situations that make them unable to receive interventions;
* Refuse to provide informed consent;

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 376 (Estimated)
Dates: Start 2022-08-01 (Estimated); Primary Completion 2025-08-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline Cardiovascular risk (Framingham risk score (FRS)) at 1 year. | Baseline; 1 year
  Cardiovascular risk is assessed by "Framingham risk score (FRS)". (Circulation, 2008,117(6): 743-753.) Generally, the "Framingham risk score (FRS)" ranges from -4 to 33 for men and -5 to 33 for women. A higher "Framingham risk score (FRS)" means a higher risk of developing cardiovascular disease.

SECONDARY OUTCOMES:
Change from baseline systolic blood pressure at 1 year after enrollment. | Baseline; 1 year
Change from baseline diastolic blood pressure at 1 year after enrollment. | Baseline; 1 year
Change from baseline fasting blood glucose at 1 year after enrollment. | Baseline; 1 year
Change from baseline glycosylated hemoglobin at 1 year after enrollment. | Baseline; 1 year
Change from baseline total cholesterol at 1 year after enrollment. | Baseline; 1 year
Change from baseline triglyceride at 1 year after enrollment. | Baseline; 1 year
Change from baseline low-density lipoprotein cholesterol at 1 year after enrollment. | Baseline; 1 year
Change from baseline high-density lipoprotein cholesterol at 1 year after enrollment. | Baseline; 1 year
Change from baseline high sensitivity C-reactive protein at 1 year after enrollment. | Baseline; 1 year
Change from baseline interleukin-6 at 1 year after enrollment. | Baseline; 1 year
Change from baseline cardiovascular risk (CHINA-PAR) at 1 year after enrollment. | Baseline; 1 year
  China-PAR is an abbreviation of "Prediction for ASCVD Risk in China". It is a prediction model developed by YANG X. (Circulation, 2016,134(19):1430-1440.) Through China-PAR, the investigators can assess one's cardiovascular risk in 10 years. The result of China-PAR is directly one's predicted cardiovascular risk in 10 years, ranging from 0% - 100%, with a higher probability meaning a higher risk of cardiovascular disease.
Change from baseline community periodontal index at 1 year after enrollment. | Baseline; 1 year
  Community periodontal index will be evaluated according to the guidelines by stomatologists. The community periodontal index ranges from 0 - 4 points for each tooth. Higher points mean more severe periodontitis.
Major adverse cardiovascular event | Baseline; 3 months; 6 months; 9 months; 1 year; 2 years; 3 years;
  The major adverse cardiovascular event includes acute myocardial infarction, stroke, heart failure, peripheral artery disease, and coronary heart disease.
All-cause mortality | Baseline; 3 months; 6 months; 9 months; 1 year; 2 years; 3 years;
  Defined as any death after enrollment.
Change from baseline anxiety at 1 year after enrollment. | Baseline; 1 year
  Anxiety will be assessed through "Self-Rating Anxiety Scale (SAS)". The SAS score range from 20 - 80 points. Higher points mean more serious anxiety.
Change from baseline pain at 1 year after enrollment. | Baseline; 1 year
  The degree of pain will be assessed through "Visual Analogue Scale (VAS)". The VAS score range from 0 - 10 points. Higher points mean more serious pain.

CONTACTS AND LOCATIONS:
Overall Officials: Jiancheng Xiu, MD, Principal Investigator — Nanfang Hospital, Southern Medical University
Locations (2):
- China (2):
  - Stomatological Hospital, Southern Medical University, Guangzhou, Guangdong
  - Nanfang Hospital, Southern Medical University, Guangzhou, Guangdong

IPD SHARING:
Plan to Share IPD: No